CLINICAL TRIAL: NCT06536959
Title: A Study of VA Combined With PD-1 Inhibitor in the Treatment of Relapsed and Refractory AML and High-risk MDS
Brief Title: VA Combined With PD-1 Inhibitor for the Treatment of Relapsed and Refractory AML and High-risk MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Ning Gao, Chief Physician, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA-PD1-MN
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Myelodysplastic Syndromes; Minimal Residual Disease
Keywords: Venetoclax; Hypomethylation agen; PD-1 inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasm, Residual | interventions — Immune Checkpoint Inhibitors; venetoclax; Decitabine; Azacitidine; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VA-PD1i (Experimental): Patients are treated with PD-1 inhibitor combined with venetoclax and decitabine/azacytidine.
  Interventions: Drug: PD-1 inhibitor, Venetoclax, Decitabine, Azacytidine

INTERVENTIONS:
Drug: PD-1 inhibitor, Venetoclax, Decitabine, Azacytidine — For AML patients: PD-1 inhibitor was given at a dose of 200mg on day 21 of the treatment. Venetoclax was given at a dose of 400 mg/day for 28 days per cycle. Decitabine was given at a dose of 20 mg/m2/day for 5 days or azacytidine was given at a dose of 75 mg/m2/day for 7 days at the discretion of the treating physician.
  For MDS patients: PD-1 inhibitor was given at a dose of 200mg on day 21 of the treatment. Venetoclax was given at a dose of 400 mg/day for 14 days per cycle. Decitabine was given at a dose of 20 mg/m2/day for 5 days or azacytidine was given at a dose of 75 mg/m2/day for 7 days at the discretion of the treating physician.
  The venetoclax starting dose is 100 mg on the first day, ramping up to 200 mg on the second day and finally 400 mg once daily. The steady daily dose (after ramp-up phase) should be reduced to 100 mg (coadministered with moderate CYP3A inhibitors or P-gp inhibitors) and 70 mg (coadministered with strong CYP3A4 inhibitors).
  Other Names: PD-1 inhibitor (Tislelizumab); Venetoclax (ABT-199, GDC-0199); Decitabine (Dacogen, 5-aza-2-deoxycytidine); Azacitidine (5-Azacytidine, Ladakamycin)

SUMMARY:
The efficiency and safety of PD-1 inhibitor in combination with venetoclax and hypomethylation agent in relapsed/refractory acute myeloid leukemia or high-risk myelodysplastic syndrome remain uncertain. In this study, the investigators aimed to assess safety and response to a new PD-1 inhibitor-based triple-drug combination regimen (venetoclax + hypomethylation agent + PD-1 inhibitor) in relapsed/refractory acute myeloid leukemia and high-risk myelodysplastic syndrome patients, or who had positive minimal residual disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with relapsed and refractory acute myeloid leukemia (AML) and patients diagnosed with myelodysplastic syndrome (MDS) who require chemotherapy treatment.
* Patients who did not respond or had disease recurrence after 1 course of induction chemotherapy or had positive immune residues after induction chemotherapy or positive molecular residues (if any) after induction chemotherapy.
* Voluntarily participate in clinical research and sign an informed consent form and be willing to follow and be able to complete all experimental procedures.
* The toxic and side effects caused by the last treatment should be recovered.
* Eastern Cooperative Oncology Group score of 0 to 3 points.
* The organ function is intact.

  * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2×ULN (Upper Limit of Normal).
  * Creatinine≤2×ULN.
  * Bilirubin≤2×ULN.
* Karnofsky≥70.
* The expected survival period is at least 12 weeks.
* Non-pregnant, non-breastfeeding women.

Exclusion Criteria:

* Suffering from other untreated or unrelieved malignant tumors within 2 years.
* Major surgery, radiotherapy, chemotherapy, biological therapy, immunotherapy, and experimental therapy were performed within 2 weeks of the first medication.
* Suffering from any other known serious and/or uncontrolled disease (eg, uncontrolled diabetes; cardiovascular disease, including congestive heart failure New York Heart Association [NYHA] Class III or IV, 6 months patients with myocardial infarction and poorly controlled blood pressure); chronic renal failure; or active uncontrolled infection); the investigators considered unsuitable for this clinical trial.
* Patients who are unwilling or unable to comply with the protocol.
* Currently being treated with other systemic anti-tumor or anti-tumor research drugs.
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | At the end of Cycle 2 (each cycle is 28 days)
  percentage of subjects with complete remission (CR) and incomplete hematologic recovery (CRi)
Complete minimal residual disease (MRD) Response Rate | At the end of Cycle 2 (each cycle is 28 days)
  Percentage of subjects with MRD negative or MRD < 0.01%
MRD Response Rate | At the end of Cycle 2 (each cycle is 28 days)
  Percentage of subjects with MRD < 0.1% detectable by multicolor flow cytometry

SECONDARY OUTCOMES:
Relapse-Free Survival | 24 months
  Time interval from leukemia free state to the first recurrence or death
Overall Survival | 24 months
  Time interval from start of treatment until death or last follow-up
Duration of response | 24 months
  Time interval from morphologic/MRD response to loss of response or death
Adverse events | start of treatment to 2 weeks after end of treatment
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao-ning Gao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No